CLINICAL TRIAL: NCT05101967
Title: Dynamic Cervical Implant (DCI) vs. Anterior Cervical Discectomy and Fusion (ACDF) in Treatment of Single-level Cervical Disc Prolapse
Brief Title: Dynamic Cervical Implant vs. Anterior Cervical Discectomy and Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, H A Othman, Registrar, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCI vs. ACDF
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cervical Disc Prolapse
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Cervical Implant (Experimental)
  Interventions: Procedure: Dynamic Cervical Implant
- Anterior Cervical Discectomt and Fusion (Active Comparator)
  Interventions: Procedure: Anterior Cervical Discectomt and Fusion

INTERVENTIONS:
Procedure: Dynamic Cervical Implant — Cervical discectomy through anterior approach with replacement of disc by dynamic implant
  Arms: Dynamic Cervical Implant
Procedure: Anterior Cervical Discectomt and Fusion — Cervical discectomy through anterior approach with putting of cervical cage.
  Arms: Anterior Cervical Discectomt and Fusion

SUMMARY:
Comparison between Dynamic Cervical Implant as a recently introduced technique in our department and the conventional Anterior Cervical Discectomy and Fusion in management of single-level cervical disc prolapse.

DETAILED DESCRIPTION:
Anterior cervical discectomy and fusion (ACDF) is considered to be a highly successful surgical technique for cervical spondylosis associated with brachialgia and/or myelopathy. Non-union accounts for more than two-thirds of failures in ACDF surgeries and iliac bone graft morbidity is also reported in about one-third of multilevel fusion operations. There are many types of cages used to avoid the complications associated with iliac bone grafting.These problems include persistent donor-site pain, infection, hematoma formation, iliac crest fracture, and neuralgia parasthetica.

However, in spite of being successful for many years, ACDF has its own complications in the form of non-union, implant failure, and adjacent level disease which occurs due to the excessive motion observed at the levels immediately above and/or below the index level. It has been proven to provide clinical stability after decompression.. However, although it achieves long-term success, ACDF is not without complications as there have been reports of pseudoarthrosis, implant failure, and adjacent level disease which occurs due to the significant amount of increased motion observed at the levels immediately above and below the fusion. However, greater compensation occurred at the inferior segments compared to the superior segments for the lower level fusions.

Dynamic cervical Implant (DCI) is a titanium implant, originally invented in 2002 by Dr. Guy Matgé, Luxembourg. It was introduced in clinical use, in 2004. The design was modified to better accommodate the normal disc anatomy. The DCI implant with its motion preservation characters is unique implant. It stabilizes the cervical spine while still offering a limited, controlled flexion and extension movements allowing the spine to dynamically perform its function. It also acts as a shock absorber, preventing accelerated degeneration in adjacent segments. Thus, the DCI implant aims at combining the advantages of the gold standard "fusion" with a motion preservation philosophy.

This study aims to

* compare the clinical and radiographic outcomes of ACDF versus DCI in patients with degenerative cervical radiculopathy and/or myelopathy operated upon at Assiut University Hospital.
* Give the effective treatment, pain control and can detect the best method could be used in such cases.

I.

• Improve the outcome of these patients and decease rate of recurrence and complications

ELIGIBILITY:
Inclusion Criteria:

1. Patients with single level cervical disc prolapse in the subaxial cervical vertebrae (C3 - C7) confirmed by MRI.
2. Age of the patient is between 18- 60 years old of both sex.
3. Patients are fit for surgery..

Exclusion Criteria:

1. Patients with multilevel cervical disc prolapse.
2. Patients with recurrent disc prolapse.
3. Spinal deformity
4. Spinal instability.
5. Patients who are unfit for surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of neck pain | six months
  Subjective Neck pain intensity on scale of 1-10
Visual Analogue Scale (VAS) of brachialgia | six months
  Subjective brachialgia intensity on scale of 1-10
Intervertebral Hight | six months
  The distance from the midpoint of the upper endplate of the upper vertebral body to the midpoint of the lower endplate of the lower vertebral body
Range of motion | six months
  range of motion of affected level using Cobb's angle.

SECONDARY OUTCOMES:
Blood Loss | immediate post operative
  intraoperative blood loss
Hospital Stay | up to one week
  post operative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Abokresha, Professor, Study Chair — Assiut University; Shady A Hassaan, MD, Study Director — Assiut University; Hazem A Othman, MSc, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No